CLINICAL TRIAL: NCT03002194
Title: Change in Skin Elasticity After Combined Radiofrequency and Electromagnetic Treatment
Brief Title: Change in Skin Elasticity With RF and PEMF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0316
Record Dates: First submitted 2016-11-24; First posted 2016-12-23 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Skin Abnormalities
Keywords: rhytides; wrinkle
MeSH Terms: conditions — Skin Abnormalities | interventions — Moire Topography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RF and PEMF therapy (Experimental): Each subject is to receive 8 weekly study treatments. The study treatment consists of Glide (medical grade glycerin) being applied thoroughly to the study treatment area (face). The energy will be delivered by the Diamondpolar applicator attached to the Venus Versa, a medical device approved by health regulatory authorities, to deliver combined radiofrequency (RF) and pulsed electromagnetic field (PEMF) energies. Change in skin elasticity will be measured by Cutometer. Change in appearance will be assessed by independent reviewer using photographs.
  Interventions: Device: Cutometer; Other: Photographs

INTERVENTIONS:
Device: Cutometer — Skin elasticity will be measured by a Cutometer prior to beginning treatment, week 7 and 3 months after completion of the treatment.
Other: Photographs — Photographs will be taken prior to beginning treatment, week 7 and 3 months after completion of the treatment.

SUMMARY:
This study will measure the difference in skin elasticity in females only before and after treatment with radiofrequency and pulsed electromagnetic field therapy.

DETAILED DESCRIPTION:
This study is an open-label, baseline-controlled, single-center study to measure the change in skin elasticity after combined radio frequency (RF) and pulsed electromagnetic field (PEMF) treatment. Forty-five adult females will undergo weekly treatments over a period of 8 weeks. Skin elasticity will be measured by a Cutometer® prior to beginning treatment, week 7 and 3 months after completion of treatment. Photographs will be taken prior to treatment, at week 4, week 7 and 3 months after completion of treatment. Patient discomfort/pain and satisfaction questionnaires will be completed before, during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult female subject, 18 years of age and older with Fitzpatrick skin types I-IV
* Ability to tolerate the RF/PEMF procedure, and willing to adhere to the treatment regimen

Exclusion Criteria:

* Having any active electrical implant or permanent implant anywhere in the body, e.g. pacemaker, internal defibrillator
* Prior use of retinoids in treated area within 2 weeks of initial treatment
* Use of oral Isotretinoin (Accutane®) within 6 months of initial treatment
* Patient on systemic corticosteroid therapy 6 months prior to start of study
* Prior use of collagen, fat injections and /or other methods of skin augmentation (enhancement with injected or implanted material) in treated area within 4-6 weeks of initial treatment. Treatment may not be performed at all over permanent dermal implants.
* Prior ablative resurfacing procedure in treated area with laser or other devices within 12 months of initial treatment
* Any other surgery in treated area within 12 months of initial treatment
* History of keloid formation or poor wound healing in a previously injured skin area
* Epidermal or dermal disorders
* Open laceration or abrasion of any sort on the area to be treated.
* History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or use of immunosuppressive medications.
* Having any form of active cancer at the time of enrollment
* Significant concurrent illness, such as uncontrolled diabetes i.e. any disease state that in the opinion of the Investigator would interfere with the treatment, or healing process
* Participation in a study of another device or drug within 1 month prior to study enrollment
* Tattoos in the treatment area.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoni Iger, PhD, Study Director — Venus Concept Ltd.
Locations (1):
- Art of Facial Surgery, North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RF and PEMF Therapy
Started | 48
Completed | 38
Not Completed | 10
Not completed — Lost to Follow-up | 6
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group: Each subject is to receive 8 weekly study treatments. The study treatment consists of Glide (medical grade glycerin) being applied thoroughly to the study treatment area (face). The energy will be delivered by the Diamondpolar applicator attached to the Venus Versa, a medical device approved by health regulatory authorities, to deliver combined radiofrequency (RF) and pulsed electromagnetic field (PEMF) energies.
Arm/Group | Treatment Group
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 10
Sex/Gender, Customized [Number; unit: participants]
  Female | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 43
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  Canada | 48
Baseline cutometer reading [Mean (Standard Deviation); unit: ratio] — Change in skin elasticity will be measured by a Cutometer prior to beginning treatment. The ratio R2 describes the change in gross elasticity as a ratio of maximum recovery (Ua) and skin distensibility (Uf) (Ua/Uf).
  ratio | 0.7658 (0.1127)

OUTCOME MEASURES:

1. Primary Outcome: Change in Facial Skin Elasticity
Description: A Cutometer® will be used to measure the change in gross elasticity (R2) of the facial skin as calculated by Ua/Uf which is a ratio of maximum recovery (Ua) and skin distensibility (Uf). The value is expressed as a percentage, the closer the value is to 1 (100%), the more elastic the skin.
Time Frame: 20 weeks after the last study treatment
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | RF and PEMF Therapy
Number analyzed (Participants) | 38
ratio
  Mean R2 Cutometer Reading Baseline | 0.7658 (0.1127)
  Mean R2 Cutometer Reading Wk 20 | 0.7244 (0.1487)

2. Secondary Outcome: Improvement in Subject Satisfaction With Facial Skin Laxity Compared to Baseline as Measured by the 5-point Likert Satisfaction Scale
Description: Subject will assign a score that best represents the level of satisfaction they have in their appearance as a result of the study treatment. The scale reports five categories - 4 - very satisfied; 3 - satisfied; 2 - having no opinion; 1 - unsatisfied and 0 - very unsatisfied. The higher the score, the more satisfaction with the treatment that a subject reports.
Time Frame: 7 weeks and 20 weeks post study treatments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RF and PEMF Therapy
Number analyzed (Participants) | 38
score on a scale
  Mean Satisfaction week 7 post Tx | 3.11 (0.92)
  Mean Satisfaction Week 20 post Tx | 2.58 (1.12)

3. Secondary Outcome: General Aesthetic Improvement Scale (GAIS)
Description: Subject to assess their general improvement in appearance at 7 and 20 weeks post-intervention using a 7 category scale: 3 - very much improved; 2 - much improved; 1 - improved; 0 - no change; -1 - worse; -2 - much worse and -3 very much worse. The higher the positive score, the more the subject feels their appearance has changed for the better.
Time Frame: 7 weeks and 20 weeks post study treatments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RF and PEMF Therapy
Number analyzed (Participants) | 38
score on a scale
  Mean GAIS week 7 post Tx | 1.19 (0.92)
  Mean GAIS week 20 post Tx | 0.58 (0.74)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 9 months and 18 days. All reportable events with start dates occurring any time after informed consent is obtained will be followed until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation.
Arm/Group | RF and PEMF Therapy
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT03002194/Prot_SAP_000.pdf